CLINICAL TRIAL: NCT03244800
Title: A Phase 2, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Different Doses of MEDI0382 in Overweight and Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Investigate Different Doses of 0382 in Overweight and Obese Subjects With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5670C00011
Record Dates: First submitted 2017-07-27; First posted 2017-08-10 (Actual); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: 0382, T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Cohort 1 (Placebo Comparator): Participants will receive placebo matching with MEDI0382 subcutaneously once daily for 49 days.
  Interventions: Drug: Placebo
- MEDI0382 Cohort 1 (Experimental): Participants will receive subcutaneous injection of MEDI0382 once daily for 49 days as Dose 1 for 7 days, followed by Dose 2 for 7 days, Dose 3 for 7 days, and Dose 4 for 28 days
  Interventions: Drug: MEDI0382
- PLacebo Cohort 2 (Placebo Comparator): Participants will receive placebo matching with MEDI0382 subcutaneously once daily for 49 days.
  Interventions: Drug: Placebo
- MEDI0382 Cohort 2 (Experimental): Participants will receive subcutaneous injection of MEDI0382 once daily for 49 days as Dose 1 for 14 days, followed by Dose 2 for 14 days, Dose 3 for 14 days, and Dose 4 for 7 days.
  Interventions: Drug: MEDI0382

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 will be administered subcutaneously once daily for 49 days.
  Arms: MEDI0382 Cohort 1; MEDI0382 Cohort 2
Drug: Placebo — Placebo will be administered subcutaneously once daily for 49 days.
  Arms: PLacebo Cohort 2; Placebo Cohort 1

SUMMARY:
A Phase 2 study with two cohorts of differing doses designed to evaluate the efficacy, safety and pharmacokinetics (PK) of MEDI0382 in patients with Type 2 Diabetes Mellitus (T2DM). Approximately 63 subjects will be enrolled across two cohorts.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled study designed to evaluate the efficacy, safety, tolerability, and pharmacokinetics of different doses of MEDI0382 administered as multiple SC doses to subjects with T2DM. Approximately 63 subjects will be enrolled across two cohorts.

For cohort 1, sufficient subjects will be invited to participate in the study such that a maximum of 39 subjects will complete dosing. Subjects in cohort 1 will be randomised using a ratio of 2:1 to one of 2 treatment arms to receive either MEDI0382 or placebo. A maximum of 26 will complete dosing in the active arm and 13 will complete dosing in the placebo arm.

For cohort 2, sufficient subjects will be invited to participate in the study such that a maximum of 24 subjects will complete dosing. Subjects in cohort 2 will be randomised using a ratio of 3:1 to receive either MEDI0382 or placebo. A maximum of 18 will complete dosing in the active arm and 6 will complete dosing in the placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged ≥ 18 years at screening
2. Provision of signed and dated written informed consent
3. BMI between 27 and 40 kg/m2
4. HbA1c range of 6.5% to 8.5%
5. Diagnosed with T2DM with glucose control managed with metformin monotherapy where no significant dose change (increase or decrease ≥ 500 mg/day) has occurred in the 3 months prior to screening
6. Subjects prescribed oral dual therapy with a dipeptidyl peptidase-4 inhibitor, sulphonylurea, glitinide, or a sodium-glucose co-transporter 2 inhibitor in addition to metformin at screening may be eligible to enter the study following a 4-week washout period
7. Female subjects of childbearing potential must have a negative pregnancy test at screening and randomisation, and must not be lactating
8. Females of childbearing potential who are sexually active with a nonsterilised male partner must use at least one highly effective method of contraception from screening and must agree to continue using such precautions through to the end of the study. It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

1. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product, put the subject at risk, influence the subject's ability to participate or affect the interpretation of the results of the study and/or any subject unable or unwilling to follow study procedures
2. Concurrent participation in another study of any kind and repeat randomisation in this study is prohibited
3. Severe allergy/hypersensitivity to any of the proposed study treatments
4. Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus or diabetic ketoacidosis, or if the subject has been treated with daily SC insulin within 90 days prior to screening
5. Significant inflammatory bowel disease, gastroparesis, or other severe disease or surgery affecting the upper GI tract (including weight-reducing surgery and procedures) which may affect gastric emptying or could affect the interpretation of safety and tolerability data
6. Significant hepatic disease (except for non-alcoholic steatohepatitis or non-alcoholic fatty liver disease without portal hypertension or cirrhosis) and/or subjects with any of the following results at screening:

   * Aspartate transaminase (AST) ≥ 3 × upper limit of normal (ULN)
   * Alanine transaminase (ALT) ≥ 3 × ULN
   * Total bilirubin ≥ 2 × ULN
7. Impaired renal function defined as estimated glomerular filtration rate (GFR) < 60 mL/minute/1.73 m2 at screening (GFR estimated according to Modification of Diet in Renal Disease [MDRD] using the isotope dilution mass spectrometry [IDMS] traceable MDRD Study Equation [SI units])
8. Poorly controlled hypertension defined as:

   * Systolic BP > 160 mm Hg
   * Diastolic BP ≥ 95 mm Hg after 10 minutes of seated rest and confirmed by repeated measurement at screening.
9. Unstable angina pectoris, myocardial infarction, transient ischemic attack or stroke within 3 months prior to screening, or subjects who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
10. Severe congestive heart failure (New York Heart Association Class III or IV)
11. Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia
12. Haemoglobinopathy, haemolytic anemia, or chronic anaemia (haemoglobin concentration < 11.5 g/dL [115 g/L] for males, < 10.5 g/dL [105 g/L] for females) at screening or any other condition known to interfere with interpretation of HbA1c measurement
13. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer
14. Any positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, and human immunodeficiency virus (HIV) antibody
15. History of substance dependence, alcohol abuse, or excessive alcohol intake (defined as an average weekly intake of > 21 alcoholic drinks for men or > 10 alcoholic drinks for women) within 3 years prior to screening, and/or a positive screen for drugs of abuse or alcohol at screening or on admission to the study unit. Subjects who use tricyclic antidepressants or benzodiazepines for an established clinical indication may be permitted to enter the study based upon the judgement of the investigator.
16. Involvement of any AstraZeneca, MedImmune, contract research organization, or study site employee or their close relatives
17. History of acute or chronic pancreatitis or other diseases of the pancreas

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (5):
- Germany (5):
  - Research Site, Berlin
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Neu-Ulm
  - Research Site, Neuss

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker VER, Robertson D, Wang T, Hornigold DC, Petrone M, Cooper AT, Posch MG, Heise T, Plum-Moerschel L, Schlichthaar H, Klaus B, Ambery PD, Meier JJ, Hirshberg B. Efficacy, Safety, and Mechanistic Insights of Cotadutide, a Dual Receptor Glucagon-Like Peptide-1 and Glucagon Agonist. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz047. doi: 10.1210/clinem/dgz047. PMID 31608926
- See also: D5670C00011_protocol_amendment_2_ct — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14682&filename=D5670C00011_protocol_amendment_2_ct.pdf
- See also: D5670C00011_Statistical_Analysis_Plan — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14682&filename=D5670C00011_Statistical_Analysis_Plan.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 5 sites in Germany between 04Sep2017 and 23Jan2018.
Pre-assignment Details: A total of 120 participants consented to participate in the study. Of which 55 were screen failures; 65 participants were randomised (46 to MEDI0382 and 19 to placebo).
Groups:
- Placebo Cohort 1: Participants received placebo matching with MEDI0382 subcutaneously (SC) once daily for 49 days.
- MEDI0382 Cohort 1: Participants received subcutaneous injection of MEDI0382 once daily for 49 days as Dose 1 for 7 days, followed by Dose 2 for 7 days, Dose 3 for 7 days, and Dose 4 for 28 days.
- Placebo Cohort 2: Participants received placebo matching with MEDI0382 SC once daily for 49 days.
- MEDI0382 Cohort 2: Participants received subcutaneous injection of MEDI0382 once daily for 49 days as Dose 1 for 14 days, followed by Dose 2 for 14 days, Dose 3 for 14 days, and Dose 4 for 7 days.
Period: Overall Study
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Started | 13 | 26 | 6 | 20
Completed | 13 | 25 | 6 | 18
Not Completed | 0 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Withdrew treatment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they received.
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2 | TOTAL
Number analyzed (Participants) | 13 | 26 | 6 | 20 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (5.6) | 58.7 (8.5) | 60.3 (9.5) | 61.9 (6.0) | 60.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 1 | 10 | 22
  Male | 9 | 19 | 5 | 10 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 26 | 6 | 20 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native Asian | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  White | 13 | 25 | 6 | 20 | 64
  Other | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Percent Change From Baseline in Plasma Glucose Area Under the Concentration-time Curve From Time 0 to 4 Hours (AUC0-4h) by Mixed-meal Tolerance Test (MMTT) to Day 49
Description: The MMTT test involved the consumption of a standardised liquid meal within 5 minutes and timed serial blood samples obtained for the measurement of glucose and parameters related to glucose metabolism through 240 minutes after consumption of the standardised meal (with no additional food intake during this time). The percent change in the MMTT plasma glucose AUC 0-4h from the baseline (Day -1) to Day 49 is reported.
Time Frame: Zero minutes before and 15, 30, 45, 60, 90, 120, 180, and 240 minutes after consumption of the standardised liquid meal
Population: Pharmacodynamic (PD) population included all participants who received at least one dose of study drug and had at least one post-baseline MMTT PD sample or PD evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo Cohort 1: Participants received placebo matching with MEDI0382 SC once daily for 49 days.
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1
Number analyzed (Participants) | 13 | 26
Percent change | 6.32 [-0.74 to 13.38] | -21.52 [-26.51 to -16.54]
Statistical Analysis 1: Comparison: Placebo Cohort 1 vs MEDI0382 Cohort 1; Test type: Superiority; p < 0.001, ANCOVA

2. Primary Outcome: Cohort 1: Percent Change From Baseline in Body Weight to Day 50
Description: The percent change in body weight from baseline to Day 50 is reported.
Time Frame: Day 1 through Day 50
Population: Intent-to-treat (ITT) population included all participants who received any study drug and were analyzed according to their randomized treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1
Number analyzed (Participants) | 13 | 26
Percent change | -0.21 [-1.88 to 1.46] | -3.59 [-4.77 to -2.41]
Statistical Analysis 1: Comparison: Placebo Cohort 1 vs MEDI0382 Cohort 1; Test type: Superiority; p = 0.002, ANCOVA

3. Secondary Outcome: Cohort 1: Change From Baseline in Glycated Haemoglobin (HbA1c) to Day 49
Description: The change from baseline in Glycated haemoglobin (HbA1c) to Day 49 is reported.
Time Frame: Baseline (Day -1) through Day 49
Population: The ITT population included all participants who received any study drug and were analyzed according to their randomized treatment group.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1
Number analyzed (Participants) | 13 | 26
Percentage change | -0.07 [-0.27 to 0.14] | -0.67 [-0.82 to -0.53]
Statistical Analysis 1: Comparison: Placebo Cohort 1 vs MEDI0382 Cohort 1; Test type: Superiority; p < 0.001, ANCOVA

4. Secondary Outcome: Cohort 1: Change From Baseline in Fasting Plasma Glucose to Day 49
Description: The changes in the fasting plasma glucose level during the study period from baseline to Day 49 is reported.
Time Frame: Baseline (Day -1) through Day 49
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1
Number analyzed (Participants) | 13 | 26
mg/dL | -2.31 [-12.74 to 8.13] | -35.37 [-42.75 to -27.99]
Statistical Analysis 1: Comparison: Placebo Cohort 1 vs MEDI0382 Cohort 1; Test type: Superiority; p < 0.001, ANCOVA

5. Secondary Outcome: Cohort 1: Change From Baseline in Body Weight to Day 50
Description: The changes in the body weight during the study period from baseline to Day 50 is reported.
Time Frame: Day 1 through Day 50
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1
Number analyzed (Participants) | 13 | 26
Kilogram | -0.08 [-1.45 to 1.28] | -3.41 [-4.37 to -2.44]
Statistical Analysis 1: Comparison: Placebo Cohort 1 vs MEDI0382 Cohort 1; Test type: Superiority; p = 0.002, ANCOVA

6. Secondary Outcome: Cohort 1: Percentage of Participants Achieving Greater Than or Equal to 5% Body Weight Loss From Baseline to Day 50
Description: Participants achieving greater than or equal to 5% body weight loss from baseline to Day 50 is reported.
Time Frame: Day 1 through Day 50
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1
Number analyzed (Participants) | 13 | 26
Percentage of Participants | 7.7 | 42.3
Statistical Analysis 1: Comparison: Placebo Cohort 1 vs MEDI0382 Cohort 1; Test type: Superiority; p = 0.040, Regression, Logistic; Odds Ratio (OR) = 10.76, 90% CI 2-sided [1.61 to 72.03]

7. Secondary Outcome: Cohort 1 and Cohort 2: Percent Change From Baseline in MMTT Plasma Glucose AUC 0-4h to Day 7
Description: The MMTT test involved the consumption of a standardised liquid meal within 5 minutes and timed serial blood samples obtained for the measurement of glucose and parameters related to glucose metabolism through 240 minutes after consumption of the standardised meal (with no additional food intake during this time). The percent change in the MMTT plasma glucose AUC 0-4h from the baseline (Day -1) evaluation to Day 7 is reported.
Time Frame: Zero minutes before and 15, 30, 45, 60, 90, 120, 180, and 240 minutes after consumption of the standardised liquid meal
Population: The PD population included all participants who received at least one dose of study drug and had at least one post-baseline MMTT PD sample or PD evaluation. The number of participants analyzed at the specified time point for this outcome measure are reported.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 19
Percent change | -2.02 (11.70) | -27.17 (9.83) | 1.77 (23.43) | -31.80 (7.16)

8. Secondary Outcome: Cohort 1 and Cohort 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are the events between first doses of study drug through 7 to 14 days after the last dose of study drug (approximately 64 days).
Time Frame: From Day 1 through 7 to 14 days after the last dose of study drug (approximately 64 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 20
Participants
  TEAEs | 6 | 22 | 3 | 15
  TESAEs | 0 | 0 | 0 | 0

9. Secondary Outcome: Cohort 1 and Cohort 2: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Treatment-emergent adverse events observed in participants with clinically significant vital signs abnormalities are reported. Vital sign parameters included blood pressure, heart rate, body temperature, and respiration rate.
Time Frame: From Day 1 through 7 to 14 days after the last dose of study drug (approximately 64 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 20
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Cohort 1 and Cohort 2: Number of Participants With Abnormal Electrocardiogram Reported as TEAEs
Description: Treatment-emergent adverse events observed in participants with clinically significant ECG abnormalities are reported.
Time Frame: From Day 1 through 7 to 14 days after the last dose of study drug (approximately 64 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 20
Participants | 0 | 0 | 0 | 1

11. Secondary Outcome: Cohort 1 and Cohort 2: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator as medically significant was reported as an AE. Laboratory evaluations included haematology, serum chemistry, and urinalysis.
Time Frame: From Day 1 through 7 to 14 days after the last dose of study drug (approximately 64 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 20
Participants
  Thrombocytopenia | 0 | 0 | 0 | 1
  Hypoglycaemia | 0 | 1 | 0 | 1

12. Secondary Outcome: Cohort 1 and Cohort 2: Number of Participants With Injection Site Erythema
Description: The injection site reactions observed during study visits were reported. Injection site reactions included (but are not limited to) local erythema, pain, tenderness, induration, swelling, pruritus, ulceration, and pigmentation.
Time Frame: From Day 1 through 7 to 14 days after the last dose of study drug (approximately 64 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 20
Participants | 0 | 0 | 0 | 5

13. Secondary Outcome: Cohort 1: Area Under the Concentration-time Curve During the Dosing Interval (AUCt) of MEDI0382
Description: The area under the concentration-time curve during the dosing interval of MEDI0382 is reported.
Time Frame: Cohort 1: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 22 and 49
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline PK sample with a value above lower limit of quantification. The "Number Analyzed" denotes the number of participants analyzed at the specified time point for this outcome measure.
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Arm/Group | MEDI0382 Cohort 1
Number analyzed (Participants) | 26
ng*hr/mL
  Day 22: number analyzed (Participants) | 18
  Day 22 | 226.31 [103.95 to 488.98]
  Day 49: number analyzed (Participants) | 24
  Day 49 | 248.83 [86.57 to 558.57]

14. Secondary Outcome: Cohort 2: Area Under the Concentration-time Curve During the Dosing Interval (AUCt) of MEDI0382
Description: The area under the concentration-time curve during the dosing interval of MEDI0382 is reported.
Time Frame: Cohort 2: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 1, 7, and 14
Population: The PK population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline PK sample with a value above lower limit of quantification. The "Number Analyzed" denotes the number of participants analyzed at the specified time point for this outcome measure.
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Arm/Group | MEDI0382 Cohort 2
Number analyzed (Participants) | 20
ng*hr/mL
  Day 1: number analyzed (Participants) | 8
  Day 1 | 38.67 [34.05 to 47.25]
  Day 7: number analyzed (Participants) | 13
  Day 7 | 37.51 [8.99 to 69.82]
  Day 14: number analyzed (Participants) | 15
  Day 14 | 46.75 [26.38 to 65.61]

15. Secondary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of MEDI0382
Description: The maximum observed concentration of MEDI0382 is reported.
Time Frame: Cohort 1: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 22 and 49
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382 Cohort 1
Number analyzed (Participants) | 26
ng/mL
  Day 22: number analyzed (Participants) | 25
  Day 22 | 13.24 [4.89 to 30.3]
  Day 49: number analyzed (Participants) | 24
  Day 49 | 14.8 [5.76 to 33.3]

16. Secondary Outcome: Cohort 2: Maximum Observed Concentration (Cmax) of MEDI0382
Description: The maximum observed concentration of MEDI0382 is reported.
Time Frame: Cohort 2: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 1, 7, and 14
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382 Cohort 2
Number analyzed (Participants) | 20
ng/mL
  Day 1 | 2.00 [1.09 to 3.25]
  Day 7 | 2.53 [0.85 to 4.14]
  Day 14: number analyzed (Participants) | 19
  Day 14 | 2.65 [1.50 to 3.77]

17. Secondary Outcome: Cohort 1: Time to Reach Maximum Observed Concentration (Tmax) of MEDI0382
Description: The time to reach the maximum observed concentration of MEDI0382 is reported.
Time Frame: Cohort 1: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 22 and 49
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | MEDI0382 Cohort 1
Number analyzed (Participants) | 26
Hours
  Day 22: number analyzed (Participants) | 25
  Day 22 | 6 [4 to 12]
  Day 49: number analyzed (Participants) | 24
  Day 49 | 4 [2 to 8]

18. Secondary Outcome: Cohort 2: Time to Reach Maximum Observed Concentration (Tmax) of MEDI0382
Description: The time to reach the maximum observed concentration of MEDI0382 is reported.
Time Frame: Cohort 2: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 1, 7, and 14
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | MEDI0382 Cohort 2
Number analyzed (Participants) | 20
Hours
  Day 1 | 8 [4 to 12]
  Day 7 | 6 [0 to 8]
  Day 14: number analyzed (Participants) | 19
  Day 14 | 6 [4 to 12]

19. Secondary Outcome: Cohort 1: Terminal Half Life (t1/2) of MEDI0382
Description: The t1/2 is the time measured for the concentration to decrease by one half after the dose of MEDI0382.
Time Frame: Cohort 1: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 22 and 49
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | MEDI0382 Cohort 1
Number analyzed (Participants) | 6
Hours
  Day 22: number analyzed (Participants) | 1
  Day 22 | 9.67 [9.67 to 9.67]
  Day 49: number analyzed (Participants) | 5
  Day 49 | 8.4 [7.7 to 9.4]

20. Secondary Outcome: Cohort 2: Terminal Half Life (t1/2) of MEDI0382
Description: The t1/2 is the time measured for the concentration to decrease by one half after the dose of MEDI0382.
Time Frame: Cohort 2: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 1, 7, and 14
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: Hours
Arm/Group | MEDI0382 Cohort 2
Number analyzed (Participants) | 5
Hours
  Day 1: number analyzed (Participants) | 3
  Day 1 | 9.7 [8.9 to 10.2]
  Day 7: number analyzed (Participants) | 3
  Day 7 | 8.8 [8.6 to 9.0]
  Day 14: number analyzed (Participants) | 4
  Day 14 | 9.4 [8.7 to 10.5]

21. Secondary Outcome: Cohort 1: Accumulation Ratio (Racc) of MEDI0382
Description: The Racc was calculated using the AUC method which account for the overall exposure measured using the specified time points on Day 22 and Day 49. Racc was calculated using the formula, Racc of Day 49 = AUCt of Day 49/AUCt of Day 22.
Time Frame: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 22 and 49
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | MEDI0382 Cohort 1
Number analyzed (Participants) | 21
Ratio | 1.46 [1.13 to 2.98]

22. Secondary Outcome: Cohort 2: Accumulation Ratio of MEDI0382
Description: The Racc was calculated using the AUC method which account for the overall exposure measured using the specified time points on Day 1, Day 7 and Day 14. Racc was calculated using the formulas: Racc of Day 7 = AUCt of Day 7/AUCt of Day 1; Racc of Day 14 = AUCt of Day 14/AUCt of Day 1.
Time Frame: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 1, 7, and 14
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | MEDI0382 Cohort 2
Number analyzed (Participants) | 20
Ratio
  Day 7: number analyzed (Participants) | 13
  Day 7 | 1.36 [1.2 to 1.6]
  Day 14: number analyzed (Participants) | 13
  Day 14 | 1.46 [1.2 to 1.9]

23. Secondary Outcome: Cohort 1: Trough Plasma Concentration (Ctrough) of MEDI0382
Description: Trough plasma concentration is the measured concentration from the plasma concentration-time data at the end of a dosing interval at steady state.
Time Frame: Cohort 1: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 22 and 49
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382 Cohort 1
Number analyzed (Participants) | 26
ng/mL
  Day 22: number analyzed (Participants) | 25
  Day 22 | 3.566 [0.50 to 9.27]
  Day 49: number analyzed (Participants) | 24
  Day 49 | 5.762 [1.53 to 11.80]

24. Secondary Outcome: Cohort 2: Trough Plasma Concentration (Ctrough) of MEDI0382
Description: Trough plasma concentration is the measured concentration from the plasma concentration time data at the end of a dosing interval at steady state.
Time Frame: Cohort 2: Predose and 1, 2, 4, 6, 8, and 12 hours postdose on Days 1, 7, and 14
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382 Cohort 2
Number analyzed (Participants) | 20
ng/mL
  Day 1: number analyzed (Participants) | 0
  Day 7: number analyzed (Participants) | 19
  Day 7 | 1.147 [0.79 to 2.36]
  Day 14: number analyzed (Participants) | 19
  Day 14 | 1.147 [0.69 to 1.92]

25. Secondary Outcome: Cohort 1 and Cohort 2: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI0382
Description: Participants with positive serum antibodies to MEDI0382 are reported.
Time Frame: Baseline (Day 1), Day 29, Day 50, and Follow-up Visit 2 (28 days after the last dose [approximately 64 days])
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they received. The "Number Analyzed" denotes the number of participants analyzed at the specified time point for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 13 | 26 | 6 | 20
Participants
  Baseline (ADA positive) | 0 | 0 | 0 | 0
  Day 29 (ADA positive): number analyzed (Participants) | 13 | 26 | 6 | 18
  Day 29 (ADA positive) | 0 | 4 | 0 | 1
  Day 50 (ADA positive): number analyzed (Participants) | 13 | 25 | 6 | 18
  Day 50 (ADA positive) | 0 | 7 | 0 | 2
  Follow-up Visit 2 (ADA positive): number analyzed (Participants) | 13 | 24 | 6 | 20
  Follow-up Visit 2 (ADA positive) | 1 | 6 | 0 | 6

ADVERSE EVENTS:
Time Frame: From Day 1 through 7 to 14 days after the last dose of study drug (approximately 64 days)
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/26 | 0/6 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/26 | 0/6 | 0/20
Other Adverse Events (participants affected / at risk) | 6/13 | 22/26 | 3/6 | 15/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=13) | MEDI0382 Cohort 1 (N=26) | Placebo Cohort 2 (N=6) | MEDI0382 Cohort 2 (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (8) | 0 (0) | 2 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (8) | 0 (0) | 7 (11)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (6) | 0 (0) | 4 (11)
Face oedema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4) | 3 (4) | 0 (0) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 13 (17) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (6)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Loss of libido (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03244800/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03244800/SAP_001.pdf